CLINICAL TRIAL: NCT05415020
Title: Feasibility, Acceptability, and Pilot Testing of a Behavioral Intervention for Chronic Migraine
Brief Title: Determining the Utility of a Behavioral Intervention in Chronic Migraine
Acronym: RLB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Yohannes Woubishet Woldeamanuel, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-004888; K01NS124911 (NIH)
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Migraine; Headache; Migraine Disorders; Chronic Migraine; Lifestyle Factors; Headache Disorders
Keywords: Migraine Disorders; Headache; Lifestyle
MeSH Terms: conditions — Migraine Disorders; Headache; Headache Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Therapy Group (Active Comparator)
  Interventions: Behavioral: Lifestyle Behavior Protocol
- Attention Placebo Group (Sham Comparator)
  Interventions: Behavioral: Sham Behavior Protocol

INTERVENTIONS:
Behavioral: Lifestyle Behavior Protocol — Virtual training on building a skillset to improve lifestyle behavior that reduces migraine attacks
  Arms: Virtual Therapy Group
Behavioral: Sham Behavior Protocol — Virtual training on the disease of migraine and how migraine can progress to chronic migraine.
  Arms: Attention Placebo Group

SUMMARY:
This proposal will involve a pilot study to evaluate the feasibility, acceptability, and outcomes of a lifestyle behavior protocol in managing chronic migraine. Additionally, the proposal will investigate biomolecules that are uniquely involved in chronic migraine patients who respond to the protocol. Successful completion of this proposal will inform the design of a future full-scale behavioral clinical trial to control chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* have chronic migraine for a minimum of 1-year
* aged 18 years and older

Exclusion Criteria:

* other headache disorders including secondary headache disorders
* children younger than 18 years old
* current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Number of Interested Participants that are Enrolled | 12 weeks
  Recruitment rate (Feasibility Outcome)
Acceptability | 12 weeks
  Retention rate

SECONDARY OUTCOMES:
Mean change from baseline monthly migraine frequency | 12 weeks
  Change in the mean of monthly migraine frequency
Migraine severity | 12 weeks
  severity of migraine attacks rated from 0 to 10

OTHER OUTCOMES:
Headache self-efficacy | 12 weeks
  Headache self-efficacy measured using the validated Headache Self-Efficacy Questionnaire. Scores range from 25 to 175. Higher scores mean a better outcome.
Levels of candidate biomarkers | 12 weeks
  Using mass spectrometry, serum levels of candidate biomarkers acryloyl-CoA, glutaminylhistidine, HABP2 will be compared at baseline and end of study (end of week-12)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Yohannes W. Woldeamanuel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication, for 5 years
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Woldeamanuel YW, Blayney DW, Jo B, Fisher SE, Benedict C, Oakley-Girvan I, Kesler SR, Palesh O. Headache outcomes of a sleep behavioral intervention in breast cancer survivors: Secondary analysis of a randomized clinical trial. Cancer. 2021 Dec 1;127(23):4492-4503. doi: 10.1002/cncr.33844. Epub 2021 Aug 6. PMID 34357593
- [Background] Woldeamanuel YW, Sanjanwala BM, Cowan RP. Endogenous glucocorticoids may serve as biomarkers for migraine chronification. Ther Adv Chronic Dis. 2020 Jul 21;11:2040622320939793. doi: 10.1177/2040622320939793. eCollection 2020. PMID 32973989
- [Background] Woldeamanuel YW, Sanjanwala BM, Peretz AM, Cowan RP. Exploring Natural Clusters of Chronic Migraine Phenotypes: A Cross-Sectional Clinical Study. Sci Rep. 2020 Feb 18;10(1):2804. doi: 10.1038/s41598-020-59738-1. PMID 32071349
- [Background] Woldeamanuel YW, DeSouza DD, Sanjanwala BM, Cowan RP. Clinical Features Contributing to Cortical Thickness Changes in Chronic Migraine - A Pilot Study. Headache. 2019 Feb;59(2):180-191. doi: 10.1111/head.13452. Epub 2018 Nov 23. PMID 30468246
- [Background] Woldeamanuel YW, Cowan RP. Migraine affects 1 in 10 people worldwide featuring recent rise: A systematic review and meta-analysis of community-based studies involving 6 million participants. J Neurol Sci. 2017 Jan 15;372:307-315. doi: 10.1016/j.jns.2016.11.071. Epub 2016 Dec 3. PMID 28017235
- [Background] Woldeamanuel YW, Cowan RP. The impact of regular lifestyle behavior in migraine: a prevalence case-referent study. J Neurol. 2016 Apr;263(4):669-76. doi: 10.1007/s00415-016-8031-5. Epub 2016 Jan 25. PMID 26810728